CLINICAL TRIAL: NCT07138014
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Phase II Study to Evaluate the Efficacy and Safety of FHND1002 Granules in Patients With Amyotrophic Lateral Sclerosis (ALS)
Brief Title: FHND1002 for ALS Treatment: Phase 2
Acronym: FHN-ALS2
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jiangsu Chia Tai Fenghai Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FHND1002-II-01
Record Dates: First submitted 2025-08-15; First posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Amyotrophic Lateral Sclerosis (ALS)
Keywords: Amyotrophic Lateral Sclerosis (ALS); Phase II; FHND1002
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Intervention Model Description: Participants are randomized in a 1:1:1 ratio to three parallel arms:
  * Arm 1: FHND1002 100mg granules + standard ALS care
  * Arm 2: FHND1002 200mg granules + standard ALS care
  * Arm 3: Matching placebo granules + standard ALS care Stratification factors: 1) Baseline ALSFRS-R (≥40 vs <40); 2) Site of onset (limb vs bulbar).
  Double-blind treatment period: 48 weeks.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- FHND1002 100mg (Experimental): Participants receive FHND1002 granules 100mg orally once daily for 48 weeks. Administration may occur fasting or with food. Concurrent stable ALS medications (e.g., edaravone/riluzole) are permitted if maintained ≥4 weeks prior to enrollment and unchanged during the study. Standard ALS care continues throughout.
  Interventions: Drug: FHND1002 100mg
- FHND1002 200mg (Experimental): Participants receive FHND1002 granules 200mg orally once daily for 48 weeks. Administration may occur fasting or with food. Pre-existing stable ALS therapies (edaravone/riluzole) are allowed if dose-stable for ≥4 weeks pre-randomization and maintained during the trial. Standard supportive care is provided.
  Interventions: Drug: FHND1002 200mg
- Placebo (Placebo Comparator): Participants receive matching placebo granules orally once daily for 48 weeks. Administration conditions (fasting/with food) mirror active arms. Background ALS medications (edaravone/riluzole) are permitted if stabilized ≥4 weeks before enrollment and unchanged throughout the study. Standard ALS management continues.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: FHND1002 100mg — Investigational oral granules containing 100mg FHND1002 (chemical entity: 3-n-butylphthalide derivative). Administered once daily for 48 weeks. Granules are packaged in unit-dose sachets with identical appearance across all study arms. Participants dissolve contents in water prior to ingestion. Stability testing confirms compatibility with fasting or fed conditions.
  Arms: FHND1002 100mg
Drug: FHND1002 200mg — Investigational oral granules containing 200mg FHND1002 (3-n-butylphthalide derivative). Delivered as two 100mg sachets or one 200mg sachet to maintain blinding. Daily dosing regimen for 48 weeks. Granule composition matches 100mg formulation in excipients and organoleptic properties.
  Arms: FHND1002 200mg
Drug: Placebo — Placebo granules identical to active intervention in appearance, taste, packaging, and administration method. Contains inert excipients (microcrystalline cellulose, lactose monohydrate) without active
  Arms: Placebo

SUMMARY:
This is a Phase II clinical trial evaluating the effectiveness and safety of an investigational drug, FHND1002 granules, in adults with Amyotrophic Lateral Sclerosis (ALS).

The main goals are:

To determine if FHND1002 can slow the progression of ALS compared to a placebo.

To assess the safety and tolerability of two different doses of FHND1002 (100mg and 200mg) in ALS patients.

Approximately 180 participants will be randomly assigned (like flipping a coin) to one of three groups:

FHND1002 100mg once daily

FHND1002 200mg once daily

Placebo (an inactive substance) once daily Assignment will consider disease severity (ALSFRS-R score) and where symptoms started (Limb vs. Bulbar). Participants can continue taking stable doses of approved ALS medications (like riluzole or edaravone) or be on no medication.

The study consists of:

A Screening Period (up to 4 weeks).

A Double-Blind Treatment Period (48 weeks).

During the 48-week treatment period:

Participants will take their assigned granules orally once daily (with or without food).

They will attend clinic visits at Weeks 2, 4, 12, 24, 36, and 48 for safety checks.

Effectiveness will be measured at Weeks 12, 24, 36, and 48 using standard ALS assessments, including the ALS Functional Rating Scale-Revised (ALSFRS-R), breathing tests (FVC%), and quality of life/questionnaires (ROADS, ALSAQ-5).

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be ≥18 years of age at the time of signing the informed consent form.
* Subjects must have a diagnosis of Amyotrophic Lateral Sclerosis (ALS) meeting the revised El Escorial World Federation of Neurology criteria categories including Clinically Definite ALS, Clinically Probable ALS, Laboratory-supported Probable ALS, or Clinically Possible ALS.
* Subjects must demonstrate a documented mean monthly decline of ≥0.5 points in the ALS Functional Rating Scale-Revised (ALSFRS-R) score since initial diagnosis.
* During screening, subjects must exhibit a percent predicted forced vital capacity (FVC%) ≥70%; note that use of non-invasive ventilation (NIV) is exclusionary.
* Disease duration must be ≤2 years calculated from the onset of the first ALS-related symptom.
* At screening, subjects must have an ALSFRS-R total score ≥30 with a swallowing function subscore ≥2 and all respiratory-related subscores at 4 points.
* Subjects must have a Body Mass Index (BMI) ≥18.5 kg/m².
* Subjects may or may not be receiving stable therapeutic doses of approved ALS medications (e.g., edaravone, riluzole) prior to enrollment, provided any existing regimen remains unchanged throughout the study.
* Subjects must demonstrate ability to understand study procedures, willingness to comply, voluntary participation, and provide signed informed consent.

Exclusion Criteria:

* Subjects with coexisting neurological disorders that may mimic ALS symptoms or interfere with efficacy assessment (e.g., cervical/lumbar spondylosis, dementia, history of seizures except childhood febrile seizures) will be excluded.
* Subjects exhibiting motor conduction block or sensory nerve conduction abnormalities on electromyography (EMG) testing will be excluded.
* Subjects with any history of spinal surgery within 3 months prior to screening will be excluded.
* Subjects showing clinically significant laboratory abnormalities at screening including aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >1.5 × upper limit of normal (ULN), or serum creatinine (Scr) > ULN will be excluded.
* Subjects with severe/uncontrolled cardiac, hepatic, renal, hematologic, or neoplastic diseases, or active severe psychiatric disorders will be excluded.
* Exclusion applies to pregnant or lactating women, and subjects planning pregnancy during the study or within 3 months post-treatment; participants of childbearing potential unwilling to use highly effective contraception throughout the study and for 3 months after last dose are excluded.
* Subjects with known or suspected hypersensitivity to FHND1002 or its excipients will be excluded.
* Subjects who have participated in another investigational drug/device trial within 1 month prior to screening will be excluded.
* Subjects deemed by the Investigator to have any condition compromising safety, data integrity, or study compliance will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Amyotrophic Lateral Sclerosis Functional Rating Scale-Revised (ALSFRS-R) Total Score at Week 48 | Baseline to Week 48
  The difference in least-squares mean (LSMean) change from baseline to Week 48 in ALSFRS-R total score between FHND1002 treatment groups (combined or individual doses) and placebo. Missing data due to early discontinuation will be handled using multiple imputation based on observed data from the same treatment group. Analysis will use a repeated measures mixed-effects model (MMRM) adjusted for baseline ALSFRS-R score, site of onset (limb vs. bulbar), treatment group, visit, and treatment-by-visit interaction, with subject as a random effect.

IPD SHARING:
Plan to Share IPD: No
Due to privacy and confidentiality concerns, individual participant data (IPD) will not be shared. The data contains sensitive health information that is protected by regulations, and sharing it ma compromise participant confidentiality.

REFERENCES:
- [Background] Todd TW, Petrucelli L. Modelling amyotrophic lateral sclerosis in rodents. Nat Rev Neurosci. 2022 Apr;23(4):231-251. doi: 10.1038/s41583-022-00564-x. Epub 2022 Mar 8. PMID 35260846
- [Background] Fang MY, Markmiller S, Vu AQ, Javaherian A, Dowdle WE, Jolivet P, Bushway PJ, Castello NA, Baral A, Chan MY, Linsley JW, Linsley D, Mercola M, Finkbeiner S, Lecuyer E, Lewcock JW, Yeo GW. Small-Molecule Modulation of TDP-43 Recruitment to Stress Granules Prevents Persistent TDP-43 Accumulation in ALS/FTD. Neuron. 2019 Sep 4;103(5):802-819.e11. doi: 10.1016/j.neuron.2019.05.048. Epub 2019 Jul 1. PMID 31272829
- [Background] Piol D, Robberechts T, Da Cruz S. Lost in local translation: TDP-43 and FUS in axonal/neuromuscular junction maintenance and dysregulation in amyotrophic lateral sclerosis. Neuron. 2023 May 3;111(9):1355-1380. doi: 10.1016/j.neuron.2023.02.028. Epub 2023 Mar 23. PMID 36963381
- [Background] Yu CH, Davidson S, Harapas CR, Hilton JB, Mlodzianoski MJ, Laohamonthonkul P, Louis C, Low RRJ, Moecking J, De Nardo D, Balka KR, Calleja DJ, Moghaddas F, Ni E, McLean CA, Samson AL, Tyebji S, Tonkin CJ, Bye CR, Turner BJ, Pepin G, Gantier MP, Rogers KL, McArthur K, Crouch PJ, Masters SL. TDP-43 Triggers Mitochondrial DNA Release via mPTP to Activate cGAS/STING in ALS. Cell. 2020 Oct 29;183(3):636-649.e18. doi: 10.1016/j.cell.2020.09.020. Epub 2020 Oct 7. PMID 33031745
- [Background] Baughn MW, Melamed Z, Lopez-Erauskin J, Beccari MS, Ling K, Zuberi A, Presa M, Gonzalo-Gil E, Maimon R, Vazquez-Sanchez S, Chaturvedi S, Bravo-Hernandez M, Taupin V, Moore S, Artates JW, Acks E, Ndayambaje IS, Agra de Almeida Quadros AR, Jafar-Nejad P, Rigo F, Bennett CF, Lutz C, Lagier-Tourenne C, Cleveland DW. Mechanism of STMN2 cryptic splice-polyadenylation and its correction for TDP-43 proteinopathies. Science. 2023 Mar 17;379(6637):1140-1149. doi: 10.1126/science.abq5622. Epub 2023 Mar 16. PMID 36927019
- [Background] Mead RJ, Shan N, Reiser HJ, Marshall F, Shaw PJ. Amyotrophic lateral sclerosis: a neurodegenerative disorder poised for successful therapeutic translation. Nat Rev Drug Discov. 2023 Mar;22(3):185-212. doi: 10.1038/s41573-022-00612-2. Epub 2022 Dec 21. PMID 36543887
- [Background] Watanabe H, Atsuta N, Hirakawa A, Nakamura R, Nakatochi M, Ishigaki S, Iida A, Ikegawa S, Kubo M, Yokoi D, Watanabe H, Ito M, Katsuno M, Izumi Y, Morita M, Kanai K, Taniguchi A, Aiba I, Abe K, Mizoguchi K, Oda M, Kano O, Okamoto K, Kuwabara S, Hasegawa K, Imai T, Kawata A, Aoki M, Tsuji S, Nakashima K, Kaji R, Sobue G. A rapid functional decline type of amyotrophic lateral sclerosis is linked to low expression of TTN. J Neurol Neurosurg Psychiatry. 2016 Aug;87(8):851-8. doi: 10.1136/jnnp-2015-311541. Epub 2016 Jan 8. PMID 26746183
- [Background] Xu L, Liu T, Liu L, Yao X, Chen L, Fan D, Zhan S, Wang S. Global variation in prevalence and incidence of amyotrophic lateral sclerosis: a systematic review and meta-analysis. J Neurol. 2020 Apr;267(4):944-953. doi: 10.1007/s00415-019-09652-y. Epub 2019 Dec 3. PMID 31797084
- See also: Description the protocol of the study — https://www.chictr.org.cn/